CLINICAL TRIAL: NCT07342179
Title: CAR-T Immunomonitoring in Multiple Myeloma
Brief Title: CAR-T Immunomonitoring in Multiple Myeloma (CART I5M)
Acronym: CART I5M
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2025-A01924-45
Record Dates: First submitted 2025-12-01; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma (MM)
MeSH Terms: conditions — Multiple Myeloma | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Prospective interventional study with minimal risks and constraints, descriptive, exploratory, non-randomized, longitudinal, single-center, basic research aim.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental)
  Interventions: Other: Additional Bone Marrow cells and blood sampling

INTERVENTIONS:
Other: Additional Bone Marrow cells and blood sampling — Additional Bone Marrow cells and blood sampling

SUMMARY:
Multiple myeloma patients can be treated with cell therapy, which uses some of their own modified white blood cells (T lymphocytes) to target a protein (BCMA, or B-cell maturation antigen) found on the surface of the myeloma plasma cells. These modified T lymphocytes are called CAR T cells (chimeric antigen receptor T cells). The long-term persistence of these modified lymphocytes, or CAR-BCMA, is a recognized indicator of a good response to treatment. This research aims to study certain markers related to CAR-BCMA cell persistence. This research will be carried out in collaboration with the Laboratory of Ischemia Reperfusion, Metabolism and Sterile Inflammation in Transplantation (IRMETIST) INSERM unit U1313, located at the University of Poitiers. The proposed project will contribute to better patient care in the field of oncology, by identifying immunological cellular markers predictive of an effective response to anti-cancer treatments and/or immunotherapeutic targeting.

DETAILED DESCRIPTION:
Multiple myeloma data will be collected from initial diagnosis and relapses, treatments receive since initial diagnosis and the CAR-T therapy (start of CAR-T therapy, type of CAR-T, responder status). Before and up to 1 year after CART C Cells treatment, blood (7) and bone marrow (3) samples will be sent to a centralised laboratories to analyse immune cells, including CAR-BCMA cells, and measure the expression of certain proteins on their surface (CD95 and CD95L) and the serum-soluble CD95L protein.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 and over
* Patient with Multiple Myeloma according to international recommendations,
* Patient about to receive CAR-T cell therapy in accordance with the rules and authorizations in France.

Exclusion Criteria:

* Patients with severely impaired physical and/or psychological health, which, according to the investigator, may affect the participant's compliance with the study.
* Simultaneous participation in another study with an ongoing exclusion period.
* Individuals receiving enhanced protection, namely minors, pregnant and/or breastfeeding women, individuals deprived of their liberty by a judicial or administrative decision, individuals residing in a healthcare or social care facility, adults under legal guardianship, and finally, patients in emergency situations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2032-10-03 (Estimated); Study Completion 2032-10-03 (Estimated)

PRIMARY OUTCOMES:
TCF-1 transcription factor (MFI) expression level in circulating CD3+ T cells | up to 1 year
  TCF-1 transcription factor (MFI) expression level in circulating CD3+ T cells at baseline and correlation with the percentage of CAR-BCMA+ T cells at different follow-up time points up to 1 year after CAR-BCMA treatment
TCF-1 transcription factor (MFI) expression level in correlation with the depth of the patient's response as defined by international guidelines (IMS/IMWG criteria) | Up to 1 year
  TCF-1 transcription factor (MFI) expression level in correlation with the depth of the patient's response as defined by international guidelines (IMS/IMWG criteria)

SECONDARY OUTCOMES:
Stemness correlation with the persistence of CAR-BCMA lymphocytes and in the bone marrow at 3 months and 12 months after CAR-BCMA treatment | Up to 1 year
  To determine whether stemness, reflected by the expression of the transcription factor TCF1 in T lymphocytes (CD3+) before apheresis and/or lymphodepletion, is correlated with the persistence of CAR-BCMA lymphocytes in the patient, in the bone marrow at 3 months and 12 months after CAR-BCMA treatment
Expression of membrane CD95 in peripheral blood | Up to 1 year
  Identify the mechanisms of immune response homeostasis, reflected by the expression of membrane CD95L and early differentiation, interfering with the persistence of CAR-BCMA(+) T cells in peripheral blood at different time points over 12 months after CAR-BCMA treatment
Inflammatory profile of patients | Up to 1 year
  To determine whether the inflammatory profile of patients, as determined by cytokine assays (sCD95L, IL-1β, IFN-γ, IL-6, IL-10, IL-15, and TNF-α) at each time point, is inversely correlated with the persistence of CAR-BCMA(+) T cells in the periphery and/or in the bone marrow

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2025-10-28): https://cdn.clinicaltrials.gov/large-docs/79/NCT07342179/Prot_000.pdf